CLINICAL TRIAL: NCT00377364
Title: Acetaminophen for Mood and Memory Changes Associated With Prednisone Therapy
Brief Title: Acetaminophen (Tylenol) for Mood and Memory Changes Associated With Corticosteroid Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 022006-009
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Asthma; Rheumatic Disease
Keywords: Acetaminophen; corticosteroids; prednisone
MeSH Terms: conditions — Asthma; Rheumatic Diseases | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen (Experimental): Participants will be given acetaminophen (two 500 mg tablets) four times daily for 7 days.
  Interventions: Drug: Drug: Acetaminophen, Drug: Placebo
- Placebo (Placebo Comparator): Participants will be given an identical appearing placebo (two 500 mg tablets) four times daily for 7 days.
  Interventions: Drug: Drug: Acetaminophen, Drug: Placebo

INTERVENTIONS:
Drug: Drug: Acetaminophen, Drug: Placebo — Acetaminophen: Participants will be given acetaminophen (two 500 mg tablets) four times daily for 7 days, not exceeding 4,000 mg/day. Placebo: Participants will be given placebo(two 500 mg tablets) four times daily for 7 days
  Other Names: Tylenol

SUMMARY:
Studies in humans and animals support that stress and/or elevations in corticosteroids lead to changes in hippocampal structure and functioning. This is important as patients with major depression frequently have elevated cortisol, and millions of patients receive prescription corticosteroids (e.g. prednisone). Both depression and corticosteroid therapy are associated with memory impairment and hippocampal atrophy. Our research uses corticosteroid-treated patients to explore interventions that might protect the brain from the effects of stress or corticosteroids. We propose to give 30 corticosteroid-treated asthma patients acetaminophen or placebo. Between group differences in mood, memory and other neurocognitive measures will serve as outcome measures.

DETAILED DESCRIPTION:
SCIENTIFIC PROPOSAL

Aims Primary

1. Determine if patients receiving prescription corticosteroid therapy who are given acetaminophen have smaller declines in declarative memory than those receiving placebo.
2. Determine if patients receiving prescription corticosteroid therapy who are given acetaminophen have smaller increases in manic/hypomanic symptoms than those receiving placebo.

Secondary

1. Determine if patients receiving prescription corticosteroid therapy who are given acetaminophen have smaller declines in cognitive domains other than declarative memory such as working memory and executive functioning than those receiving placebo.
2. Determine if patients receiving prescription corticosteroid therapy who are given acetaminophen have smaller increases in depressive symptoms than those receiving placebo.

Background/Significance

Impact of stress or corticosteroids on the hippocampus:

Studies in animals suggest that stress-induced elevations in endogenous corticosteroids or the administration of exogenous corticosteroids are associated with cognitive deficits and changes in hippocampal structure which can (after extended exposure) include irreversible neuronal loss (Brown et al. 1999, 2004a; McEwen 1997, 2000). These findings have important implications as common psychiatric illnesses including major depressive and bipolar disorders are frequently associated with acute or chronic elevations in cortisol (Brown et al. 1999). In addition, each year approximately 10 million Americans are given prescription corticosteroids, such as prednisone or dexamethasone, for illnesses such as asthma, allergies, arthritis, and dermatological conditions (Brown et al. 1999).

The hippocampus is important as it mediates important cognitive processes and provides negative feedback to the hypothalamic-pituitary-adrenal (HPA) axis (Jacobson & Sapolsky 1991). Thus, hippocampal impairment could result in both memory loss and potentially even greater cortisol levels due to loss of normal negative feedback. This concept of hippocampal dysfunction leading to greater elevation in cortisol levels and additional hippocampal dysfunction has been termed the "glucocorticoid cascade hypothesis" (Sapolsky et al. 1986).

Several lines of evidence suggest that stress and corticosteroids may impair human hippocampal structure and functioning. Starkman et al. (1992) examined hippocampal volumes using Magnetic Resonance Imaging (MRI) in 12 patients with cortisol elevations of 1-4 years duration secondary to Cushing's disease. In three patients, hippocampal volumes fell outside the 95% confidence interval reported in the literature. Atrophy correlated with mean cortisol levels. Our group recently reported poorer performance on a declarative memory task (a measure of hippocampal functioning), smaller hippocampal volume and lower levels of N-acetyl aspartate, a putative marker of neuronal viability, in a group of 17 asthma and arthritis patients receiving long-term prednisone therapy than in a control group of similar age, education level and medical history not receiving prednisone (Brown et al 2004b).

Studies in humans also suggest smaller hippocampal volumes by Magnetic Resonance Imaging (MRI) in people with chronic or recurrent major depressive or bipolar disorders (Sheline et al. 1996; Bremner et al. 2000). Although none of these studies documented elevated cortisol levels at the time of the neuroimaging, mood disorders can be associated with an elevation in cortisol. Therefore, one explanation for these findings is hippocampal atrophy due to an excess of cortisol at some point in the illness.

Corticosteroids are associated with deficits in cognitive functioning, which may occur very rapidly after exposure and long before any changes in hippocampal structure could be detected with available imaging techniques. Thus, cognitive instruments may be a sensitive measure of early changes in the hippocampus due to corticosteroids. Declarative memory, assessed with instruments such as word lists or paragraph recall, appears to be particularly sensitive to hippocampal functioning (Squire 1992). Memory deficits have been reported in patients receiving short (days) (Naber et al. 1996, Bender et al. 1988, Newcomer et al. 1994, 1999) or long term (weeks, months or years) (Brown et al. 2004b, Keenan et al. 1996) exposures to exogenous corticosteroids.

Mood symptom with prescription corticosteroids In addition to cognitive effects, corticosteroids are also associated with changes in mood. Brief courses of prescription corticosteroids are associated primarily with manic or hypomanic symptoms (Brown et al. 2002; Naber et al. 1996) although clinically significant depressive symptoms are reported in some patients (Naber et al. 1996). Longer-term exposure to lower dosages of prednisone may be associated more strongly with depressive symptoms (Brown et al. 2004b; Keenan et al. 1996). We found lifetime prednisone-induced mood disorders in 60% of patients receiving chronic prednisone therapy (Bolanos et al. 2004).

Interventions to prevent or reverse hippocampal changes secondary to stress or corticosteroids In animal models, pharmacological interventions focusing on agents that directly reduce corticosteroid levels or reduce corticosteroid-induced elevations in serotonin or glutamate have been explored. A novel antidepressant not currently available in the U.S. for use in humans, tianeptine, appears to prevent and reverse morphological changes in the rat hippocampus during a stress paradigm (Conrad et al. 1996; Watanabe et al. 1992; Magarinos et al. 1999). An additional agent, which appears to prevent stress-induced hippocampal damage in rats, is the glutamate-release inhibitor phenytoin (Watanabe et al. 1992; Magarinos et al. 1999).

If an excess of corticosteroids is associated with memory impairment and eventual hippocampal volume loss, interventions that may prevent or reverse these changes are of great importance. Memory deficits secondary to brief (days to weeks) exposure to corticosteroids are clearly reversible with medication discontinuation. Even hippocampal changes with longer term corticosteroid exposure may be reversible. Starkman et al (1999) reported significant increases in hippocampal volumes, measured on MRI, and improvement in declarative memory in 22 patients with Cushing's disease approximately 3-18 months (mean 12 months) following successful treatment and normalization of cortisol levels. We reported on the use of lamotrigine, a glutamate release inhibitor, for 12 weeks in a group of 10 patients receiving long-term prednisone therapy (Brown et al 2003). We found statistically significant improvement in declarative memory, suggestive of a neuroprotective effect on the hippocampus, following lamotrigine therapy. We recently completed a randomized, double-blind, placebo-controlled trial of phenytoin in patients receiving prednisone therapy (Brown et al 2005). Phenytoin was associated with a significantly smaller increase in hypomanic symptom severity than placebo during the prednisone exposure. However, it appears that phenytoin, not unexpectedly, may have also been associated with some negative effects on cognition. Thus, a medication with few cognitive effects may be a better choice for use in our model system.

Interventions to prevent or reverse the mood effects of prescription corticosteroids Only two controlled clinical trials have been conducted in patients with psychiatric symptoms secondary to corticosteroids. Falk et al. (1979) reported that lithium pretreatment might attenuate corticosteroid-induced mood symptoms. While 14% of patients receiving corticotropin therapy suffered from mood symptoms, none of the patients receiving corticotropin following lithium pretreatment had a mood disturbance. As discussed above, we gave a group of adult asthma patients either phenytoin or placebo at the same time they began a course of oral prednisone therapy. The group receiving phenytoin has a significantly smaller increase in manic symptom severity than the group receiving placebo (Brown et al. 2005, see also preliminary studies section). Case reports and small open-label studies suggest that lithium and other mood stabilizers including lamotrigine, carbamazepine, gabapentin, valproic acid, traditional neuroleptics (Ahmad and Rasul, 1999) and the newer atypical agents (Brown et al. 2004c) may effectively treat or prevent corticosteroid-induced mood symptoms after their development (Brown, 2003, Brown et al. 2003).

Our group has developed a research program using humans who receive prescription corticosteroids as anti-inflammatory and immunosuppressant therapy to explore the effects of the stress hormones on the hippocampus. Our current focus is on interventions that may prevent or reverse the effects of stress or corticosteroids on the hippocampus.

Acetaminophen as a neuroprotective agent Data suggest that acetaminophen is widely distributed in the central nervous system (Caurad et al. 2001a) and may have neuroprotective properties. Pertinent to the proposed study acetaminophen protects dopaminergic neurons against glutamate excitotoxicity in vitro (Casper et al. 2000) and protects hippocampal neurons from oxidative stress (Bisaglia et al 2002). Acetaminophen also reduces staphylococcal enterotoxin-induced increases in glutamate release in the rabbit brain (Huang et al 2004). Acetaminophen also alters monoamines in the rat brain (Courad et al. 2001b), and synaptic plasticity in the hippocampus through presynaptic serotonin receptors (Chen and Bazan, 2003). No reports were found on the effect of acetaminophen on mood or memory.

Summary A reliable early effect (beginning 1-2 days into therapy) of corticosteroids on the human hippocampus is a decline in performance on declarative memory tasks (e.g. word lists). Preclinical data suggest that acetaminophen may have neuroprotective properties. We propose to give patients scheduled to receive prescription corticosteroids either acetaminophen or placebo along with the corticosteroids. Our aim is to determine if the acetaminophen attenuates the decline in declarative memory, and development of hypomanic symptomatology (e.g. insomnia, irritability, agitation) better than placebo. If this pilot study shows promising results we would anticipate conducting a larger, more definitive study, with funding from National Institutes of Health (NIH).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Scheduled to receive at least 20 mg/day of prednisone for at least 7 days
* Baseline Rey Auditory Verbal Learning Test (RAVLT) total score of ≥40

Exclusion Criteria:

* History of allergic reaction or other contraindication to acetaminophen therapy
* Acetaminophen use within 24 hours of study entry
* History of liver disease or alcohol use of greater than 3 drinks/day
* Severe or unstable medical condition (e.g., recent myocardial infarction,renal failure, diabetes with poor glycemic control)
* Pregnant or lactating female
* Patient has mental retardation, dementia, or other severe cognitive disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edson S Brown, M.D., PhD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double-blind, placebo-controlled study was conducted at asthma and allergy clinics on the UT Southwestern Medical Center campus.
Pre-assignment Details: Those with prior psychiatric symptoms during corticosteroid therapy were not excluded.
Groups:
- Acetaminophen: OTC pain reliever.fever reducer that may have neuroprotective effects.
- Placebo: Matching Placebo.
Period: Overall Study
Arm/Group | Acetaminophen | Placebo
Started | 16 | 14
Completed | 14 | 14
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (10.4) | 39.8 (11.6) | 43.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race as self reported by participants
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 8 | 18
    White | 4 | 3 | 7
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: This is a measure of declarative memory (associated with the hippocampus). The test consists of 15 nouns read aloud for five consecutive trials with each trial followed by a free-recall trial. Following the fifth trial, an interference list of 15 different words is presented followed by a free-recall trial of that list. Delayed recall of the first list is tested immediately following the interference list and after a 20-minute delay. A recognition test of 50 words including the 15 original words is presented after the delayed recall. RAVLT total score of ≥ 40 words on trials 1-5(from a range of 0 to 75 words possible)suggests relatively normal memory prior to prednisone therapy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: words
Groups:
- Acetaminophen: OTC pain reliever and fever reducer that may have neuroprotective effects.
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
words | 44.8 (4.7) | 44.1 (9.3)

2. Primary Outcome: Rey Auditory Verbal Learning Task (RAVLT)
Description: This is a measure of declarative memory (associated with the hippocampus), using the mean number of words (0-75) recalled from Trials I-V of the RAVLT ± the standard deviation. The assessement was conducted using the same procedures as at baseline. RAVLT total score of ≥ 40 words on trials 1-5(from a range of 0 to 75 words possible)suggests relatively normal memory prior to prednisone therapy.
Time Frame: Exit (Day 3 or Day 7)
Population: ITT defined as any post baseline visit. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
words | 44.9 (10.9) | 44.9 (11.2)
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Baseline RAVLT scores used as covariate; Test type: Superiority or Other; p < 0.05, ANCOVA

3. Primary Outcome: Hamilton Rating Scale for Depression (HRSD-17)
Description: The assessment is a clinician administered rating of depression with 17 questions. The total score is indicates level of depression within the following ranges: none (0-5), mild (6-10), moderate (11-15), severe (16-20), and very severe (21+).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 11.3 (6.5) | 13.4 (8.6)

4. Secondary Outcome: Internal State Scale - Activation (ISS-ACT)
Description: Activation subscale assesses (hypo)manic symptoms. There are 16 questions on the total ISS, each rated on a series of visual analogue scale (VAS) items consisting of statement followed by a 100 mm line with anchor points at 0 and 100. The 16 questions divide into four subscales measuring activation; depression, global psychopathology, and well being. Depression Index (DI): Scores for items 7 and 9 are added to give a DI score ranging from 0-200 with 0 being absence of depressive symptoms and 200 indicating severe depressive symptoms. Well-Being Index (WB): Scores for items 3, 5 and 15 are added to give a WB score ranging form 0-300, with >125 indicating euthymia. Activation Index (ACT): Scores for items 6, 8, 10, 12 and 13 are added to give an ACT score ranging from 0-500, with >155 indicating mania. Perceived Conflict Index (PC): Scores for items 1, 2, 4, 11 and 14 are added to give a PC score ranging from 0-500, with higher scores indicating greater severity of psychopathology.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 58.0 (53.8) | 109.6 (82.3)

5. Secondary Outcome: Internal State Scale - Activation (ISS-ACT)
Description: as for outcome 4
Time Frame: Exit (Day 3 or Day 7)
Population: ITT defined as any post baseline visit. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 93.5 (98.2) | 107.8 (121.0)
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA; Baseline ISS scores used as a covariate. ANCOVA results were not significant

6. Primary Outcome: Hamilton Rating Scale for Depression (HRSD-17)
Description: as for outcome 3
Time Frame: Exit (Day 3 or Day 7)
Population: ITT defined as any post baseline visit. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 8.3 (6.5) | 10.3 (8.4)
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Baseline HRSD scores used as a covariate; Test type: Superiority or Other; p < 0.05, ANCOVA

7. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: This is an 11-item, observer rated measure of the severity of manic symptoms on a 5 point scale. The total score indicates overall severity of mania with a minimum of zero (indicating normalcy) and a maximum of 60 (indicating very severe).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 5.8 (2.2) | 6.1 (5.4)

8. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 7
Time Frame: Exit (Day 3 or Day 7)
Population: ITT defined as any post baseline visit. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 5.9 (5.8) | 5.6 (5.4)
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.05, ANCOVA; Baseline YMRS scores used as a covariate

9. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: This is a seven item assessment of symptoms pertinent to asthma management, including day and nighttime symptoms; activity limitation; use of prn bronchodilators; a physiological measure of asthma (spirometry), forced expiratory volume in 1 second percent predicted (FEV1% predicted), which is the percentile of FEV1 compared to normal controls matched for age, height, gender, and race, in the scoring. Total mean is interpreted on a scale between 0 (asthma completely controlled) and 6 (asthma severely uncontrolled).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 3.1 (1.0) | 3.3 (1.3)

10. Secondary Outcome: Asthma Control Questionnaire
Description: as for outcome 9
Time Frame: Exit (Day 3 or Day 7)
Population: ITT defined as any post baseline visit. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 1.9 (1.6) | 1.7 (1.4)
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA; Baseline ACQ scores used as a covariate

ADVERSE EVENTS:
Arm/Group | Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
Limitations include the small sample size and relatively small changes in mood and memory in both groups that limited our ability to detect between-group differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No